CLINICAL TRIAL: NCT01205776
Title: Evaluation of XIENCE Versus Coronary Artery Bypass Surgery for Effectiveness of Left Main Revascularization.
Brief Title: EXCEL Clinical Trial
Acronym: EXCEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-389
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Chronic Coronary Occlusion; Unprotected Left Main Coronary Artery Disease; Stent Thrombosis; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Drug eluting stents; Stents; Unprotected Left Main Coronary Artery Disease; Coronary artery bypass graft surgery
MeSH Terms: conditions — Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous Coronary Intervention (Active Comparator): Those patients receiving the XIENCE PRIME™ EECSS or XIENCE V® EECSS or XIENCE Xpedition™ EECSS or XIENCE PRO EECSS
  Interventions: Device: Percutaneous Coronary Intervention
- Coronary Artery Bypass Graft (Active Comparator): Those patients receiving CABG
  Interventions: Procedure: CABG

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Those patients receiving the XIENCE PRIME™ EECSS or XIENCE V® EECSS or XIENCE Xpedition™ EECSS or XIENCE PRO EECSS
  Arms: Percutaneous Coronary Intervention
Procedure: CABG — Those patients receiving CABG
  Arms: Coronary Artery Bypass Graft

SUMMARY:
To establish the safety and efficacy of the commercially approved XIENCE Family Stent System (inclusive of XIENCE PRIME, XIENCE V, XIENCE Xpedition and XIENCE PRO [for use outside the United States [OUS] only]) in subjects with unprotected left main coronary artery disease by comparing to coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for RCT:

* Unprotected left main coronary artery (ULMCA) disease with angiographic diameter stenosis (DS) ≥70% requiring revascularization, or
* ULMCA disease with agniographic DS >=50% but < 70% requiring revascularization, with one or more of the following present:

  * Non-invasive evidence of ischemia referable to a hemodynamically significant left main lesion (large area of ischemia in both the LAD and LCX territories, or in either the LAD or LCX territory in the absence of other obstructive coronary artery disease to explain the LAD or LCX defect), or stress-induced hypotension or stress-induced fall in LVEF, or stress-induced transient ischemic dilatation of the left ventricle or stress-induced thallium/technetiumlung uptake, and/or
  * IVUS minimum lumen area (MLA) <= 6.0mm2, and/or
  * Fractional Flow Reserve (FFR) <=0.80
* Left Main Equivalent Disease
* Clinical and anatomic eligibility for both PCI and CABG
* Silent ischemia, stable angina, unstable angina or recent MI
* Ability to sign informed consent and comply with all study procedures including follow-up for at least three years

Exclusion Criteria:

* Clinical exclusion criteria:

* Prior PCI of the left main trunk at any time prior to randomization
* Prior PCI of any other coronary artery lesions within one year prior to randomization
* Prior CABG at any time prior to randomization
* Need for any concomitant cardiac surgery other than CABG, or intent that if the subject randomizes to surgery, any cardiac surgical procedure other than isolated CABG will be performed
* CK-MB greater than the local laboratory upper limit of normal or recent MI with CK-MB still elevated
* Subjects unable to tolerate, obtain or comply with dual antiplatelet therapy for at least one year
* Subjects requiring or who may require additional surgery within one year
* The presence of any clinical condition(s) which leads the participating interventional cardiologist to believe that clinical equipoise is not present
* The presence of any clinical condition(s) which leads the participating cardiac surgeon to believe that clinical equipoise is not present
* Pregnancy or intention to become pregnant
* Non cardiac co-morbidities with life expectancy less than 3 years
* Other investigational drug or device studies that have not reached their primary endpoint
* Vulnerable population who in the judgment of the investigator is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include: Individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention

Angiographic exclusion criteria:

* Left main diameter stenosis <50%
* SYNTAX score ≥33
* Left main reference vessel diameter <2.25 mm or >4.25 mm
* The presence of specific coronary lesion characteristics or other cardiac condition(s) which leads the participating interventional cardiologist to believe that clinical equipoise is not present
* The presence of specific coronary lesion characteristics or other cardiac condition(s) which leads the participating cardiac surgeon to believe that clinical equipoise is not present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1905 (Actual)
Dates: Start 2010-09-29 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Principal Investigator — Columbia University; Patrick W Serruys, MD, Principal Investigator — Erasmus Medical Center; Joseph Sabik, MD, Principal Investigator — Cleveland Clinical Main Campus; A. Pieter Kappetein, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

REFERENCES:
- [Derived] Giustino G, Sabik JF 3rd, Serruys PW, Puskas JD, Karmpaliotis D, Kandzari DE, Morice MC, Ragosta M 3rd, Zhang Z, Dressler O, Redfors B, Ben-Yehuda O, Sharma SK, Kappetein AP, Stone GW. Major Bleeding and Mortality After Revascularization of Left Main Disease. J Am Coll Cardiol. 2024 Dec 10;84(24):2335-2346. doi: 10.1016/j.jacc.2024.07.065. PMID 39632005
- [Derived] Ali ZA, Garcia JJ, Karimi Galougahi K, Horst J, Gallo A, Shin D, Ben-Yehuda O, Chen S, Redfors B, Kappetein AP, Sabik JF 3rd, Serruys PW, Stone GW. Impact of Incomplete Revascularization After PCI in Left Main Disease: The EXCEL Trial. Circ Cardiovasc Interv. 2024 Mar;17(3):e013192. doi: 10.1161/CIRCINTERVENTIONS.123.013192. Epub 2024 Mar 19. PMID 38502720
- [Derived] Gaba P, Sabik JF, Murphy SA, Bellavia A, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Christiansen EH, Holm NR, Nielsen PH, Sabatine MS, Stone GW, Bergmark BA. Percutaneous Coronary Intervention Versus Coronary Artery Bypass Grafting in Patients With Left Main Disease With and Without Diabetes: Findings From a Pooled Analysis of 4 Randomized Clinical Trials. Circulation. 2024 Apr 23;149(17):1328-1338. doi: 10.1161/CIRCULATIONAHA.123.065571. Epub 2024 Mar 11. PMID 38465592
- [Derived] Gaba P, Christiansen EH, Nielsen PH, Murphy SA, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Stone GW, Sabik JF, Sabatine MS, Holm NR, Bergmark BA. Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft Surgery for Left Main Disease in Patients With and Without Acute Coronary Syndromes: A Pooled Analysis of 4 Randomized Clinical Trials. JAMA Cardiol. 2023 Jul 1;8(7):631-639. doi: 10.1001/jamacardio.2023.1177. PMID 37256598
- [Derived] Magnuson EA, Chinnakondepalli K, Vilain K, Serruys PW, Sabik JF, Kappetein AP, Stone GW, Cohen DJ; EXCEL Investigators. Cost-Effectiveness of Percutaneous Coronary Intervention Versus Bypass Surgery for Patients With Left Main Disease: Results From the EXCEL Trial. Circ Cardiovasc Interv. 2022 Jul;15(7):e011981. doi: 10.1161/CIRCINTERVENTIONS.122.011981. Epub 2022 Jul 19. PMID 35861797
- [Derived] Myat A, Hildick-Smith D, de Belder AJ, Trivedi U, Crowley A, Morice MC, Kandzari DE, Lembo NJ, Brown WM III, Serruys PW, Kappetein AP, Sabik JF III, Stone G. Geographical variations in left main coronary artery revascularisation: a prespecified analysis of the EXCEL trial. EuroIntervention. 2022 Jan 28;17(13):1081-1090. doi: 10.4244/EIJ-D-21-00338. PMID 34212863
- [Derived] Gregson J, Stone GW, Ben-Yehuda O, Redfors B, Kandzari DE, Morice MC, Leon MB, Kosmidou I, Lembo NJ, Brown WM 3rd, Karmpaliotis D, Banning AP, Pomar J, Sabate M, Simonton CA, Dressler O, Kappetein AP, Sabik JF 3rd, Serruys PW, Pocock SJ. Implications of Alternative Definitions of Peri-Procedural Myocardial Infarction After Coronary Revascularization. J Am Coll Cardiol. 2020 Oct 6;76(14):1609-1621. doi: 10.1016/j.jacc.2020.08.016. PMID 33004126
- [Derived] Gaba P, Serruys PW, Sabik JF 3rd, Kappetein AP, Chen S, Morice MC, Kandzari DE, Crowley A, Mehran R, Stone GW. Effect of Baseline Anemia on Outcomes After Left Main Coronary Revascularization. J Am Coll Cardiol. 2020 Mar 31;75(12):1493-1495. doi: 10.1016/j.jacc.2020.01.037. No abstract available. PMID 32216919
- [Derived] Thuijs DJFM, Milojevic M, Stone GW, Puskas JD, Serruys PW, Sabik JF 3rd, Dressler O, Crowley A, Head SJ, Kappetein AP. Impact of left ventricular ejection fraction on clinical outcomes after left main coronary artery revascularization: results from the randomized EXCEL trial. Eur J Heart Fail. 2020 May;22(5):871-879. doi: 10.1002/ejhf.1681. Epub 2020 Feb 11. PMID 32043709
- [Derived] Giustino G, Serruys PW, Sabik JF 3rd, Mehran R, Maehara A, Puskas JD, Simonton CA, Lembo NJ, Kandzari DE, Morice MC, Taggart DP, Gershlick AH, Ragosta M 3rd, Kron IL, Liu Y, Zhang Z, McAndrew T, Dressler O, Genereux P, Ben-Yehuda O, Pocock SJ, Kappetein AP, Stone GW. Mortality After Repeat Revascularization Following PCI or CABG for Left Main Disease: The EXCEL Trial. JACC Cardiovasc Interv. 2020 Feb 10;13(3):375-387. doi: 10.1016/j.jcin.2019.09.019. Epub 2020 Jan 15. PMID 31954680
- [Derived] Kandzari DE, Gershlick AH, Serruys PW, Leon MB, Morice MC, Simonton CA, Lembo NJ, Mansour S, Sabate M, Sabik JF 3rd, Kappetein AP, Dressler O, Stone GW. Procedural characteristics and clinical outcomes in patients undergoing percutaneous coronary intervention for left main trifurcation disease: the EXCEL trial. EuroIntervention. 2020 Dec 18;16(12):e982-e988. doi: 10.4244/EIJ-D-19-00686. PMID 31793882
- [Derived] Stone GW, Kappetein AP, Sabik JF, Pocock SJ, Morice MC, Puskas J, Kandzari DE, Karmpaliotis D, Brown WM 3rd, Lembo NJ, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman PE, Bochenek A, Schampaert E, Page P, Modolo R, Gregson J, Simonton CA, Mehran R, Kosmidou I, Genereux P, Crowley A, Dressler O, Serruys PW; EXCEL Trial Investigators. Five-Year Outcomes after PCI or CABG for Left Main Coronary Disease. N Engl J Med. 2019 Nov 7;381(19):1820-1830. doi: 10.1056/NEJMoa1909406. Epub 2019 Sep 28. PMID 31562798
- [Derived] Shlofmitz E, Genereux P, Chen S, Dressler O, Ben-Yehuda O, Morice MC, Puskas JD, Taggart DP, Kandzari DE, Crowley A, Redfors B, Mehdipoor G, Kappetein AP, Sabik JF 3rd, Serruys PW, Stone GW. Left Main Coronary Artery Disease Revascularization According to the SYNTAX Score. Circ Cardiovasc Interv. 2019 Sep;12(9):e008007. doi: 10.1161/CIRCINTERVENTIONS.118.008007. Epub 2019 Sep 9. PMID 31495220
- [Derived] Thuijs DJFM, Habib RH, Head SJ, Puskas JD, Taggart DP, Stone GW, Zhang Z, Serruys PW, Sabik JF 3rd, Kappetein AP. Prognostic performance of the Society of Thoracic Surgeons risk score in patients with left main coronary artery disease undergoing revascularisation: a post hoc analysis of the EXCEL trial. EuroIntervention. 2020 May 20;16(1):36-43. doi: 10.4244/EIJ-D-19-00417. PMID 31422924
- [Derived] Modolo R, Chichareon P, Kogame N, Dressler O, Crowley A, Ben-Yehuda O, Puskas J, Banning A, Taggart DP, Kappetein AP, Sabik JA, Onuma Y, Stone GW, Serruys PW. Contemporary Outcomes Following Coronary Artery Bypass Graft Surgery for Left Main Disease. J Am Coll Cardiol. 2019 Apr 23;73(15):1877-1886. doi: 10.1016/j.jacc.2018.12.090. PMID 30999989
- [Derived] Milojevic M, Serruys PW, Sabik JF 3rd, Kandzari DE, Schampaert E, van Boven AJ, Horkay F, Ungi I, Mansour S, Banning AP, Taggart DP, Sabate M, Gershlick AH, Bochenek A, Pomar J, Lembo NJ, Noiseux N, Puskas JD, Crowley A, Kosmidou I, Mehran R, Ben-Yehuda O, Genereux P, Pocock SJ, Simonton CA, Stone GW, Kappetein AP. Bypass Surgery or Stenting for Left Main Coronary Artery Disease in Patients With Diabetes. J Am Coll Cardiol. 2019 Apr 9;73(13):1616-1628. doi: 10.1016/j.jacc.2019.01.037. PMID 30947913
- [Derived] Huang X, Redfors B, Chen S, Liu Y, Ben-Yehuda O, Puskas JD, Kandzari DE, Merkely B, Horkay F, van Boven AJ, Boonstra PW, Sabik JF, Serruys PW, Kappetein AP, Stone GW. Impact of chronic obstructive pulmonary disease on prognosis after percutaneous coronary intervention and bypass surgery for left main coronary artery disease: an analysis from the EXCEL trial. Eur J Cardiothorac Surg. 2019 Jun 1;55(6):1144-1151. doi: 10.1093/ejcts/ezy438. PMID 30596978
- [Derived] Kandzari DE, Gershlick AH, Serruys PW, Leon MB, Morice MC, Simonton CA, Lembo NJ, Banning AP, Merkely B, van Boven AJ, Ungi I, Kappetein AP, Sabik JF 3rd, Genereux P, Dressler O, Stone GW. Outcomes Among Patients Undergoing Distal Left Main Percutaneous Coronary Intervention. Circ Cardiovasc Interv. 2018 Oct;11(10):e007007. doi: 10.1161/CIRCINTERVENTIONS.118.007007. PMID 30354633
- [Derived] Giustino G, Mehran R, Serruys PW, Sabik JF 3rd, Milojevic M, Simonton CA, Puskas JD, Kandzari DE, Morice MC, Taggart DP, Gershlick AH, Genereux P, Zhang Z, McAndrew T, Redfors B, Ragosta M 3rd, Kron IL, Dressler O, Leon MB, Pocock SJ, Ben-Yehuda O, Kappetein AP, Stone GW. Left Main Revascularization With PCI or CABG in Patients With Chronic Kidney Disease: EXCEL Trial. J Am Coll Cardiol. 2018 Aug 14;72(7):754-765. doi: 10.1016/j.jacc.2018.05.057. PMID 30092952
- [Derived] Redfors B, Chen S, Crowley A, Ben-Yehuda O, Gersh BJ, Lembo NJ, Brown WM 3rd, Banning AP, Taggart DP, Serruys PW, Kappetein AP, Sabik JF 3rd, Stone GW. B-Type Natriuretic Peptide Assessment in Patients Undergoing Revascularization for Left Main Coronary Artery Disease: Analysis From the EXCEL Trial. Circulation. 2018 Jul 31;138(5):469-478. doi: 10.1161/CIRCULATIONAHA.118.033631. PMID 29666071
- [Derived] Kosmidou I, Chen S, Kappetein AP, Serruys PW, Gersh BJ, Puskas JD, Kandzari DE, Taggart DP, Morice MC, Buszman PE, Bochenek A, Schampaert E, Page P, Sabik JF 3rd, McAndrew T, Redfors B, Ben-Yehuda O, Stone GW. New-Onset Atrial Fibrillation After PCI or CABG for Left Main Disease: The EXCEL Trial. J Am Coll Cardiol. 2018 Feb 20;71(7):739-748. doi: 10.1016/j.jacc.2017.12.012. PMID 29447735
- [Derived] Baron SJ, Chinnakondepalli K, Magnuson EA, Kandzari DE, Puskas JD, Ben-Yehuda O, van Es GA, Taggart DP, Morice MC, Lembo NJ, Brown WM 3rd, Banning A, Simonton CA, Kappetein AP, Sabik JF, Serruys PW, Stone GW, Cohen DJ; EXCEL Investigators. Quality-of-Life After Everolimus-Eluting Stents or Bypass Surgery for Left-Main Disease: Results From the EXCEL Trial. J Am Coll Cardiol. 2017 Dec 26;70(25):3113-3122. doi: 10.1016/j.jacc.2017.10.036. Epub 2017 Oct 30. PMID 29097293
- [Derived] Stone GW, Sabik JF, Serruys PW, Simonton CA, Genereux P, Puskas J, Kandzari DE, Morice MC, Lembo N, Brown WM 3rd, Taggart DP, Banning A, Merkely B, Horkay F, Boonstra PW, van Boven AJ, Ungi I, Bogats G, Mansour S, Noiseux N, Sabate M, Pomar J, Hickey M, Gershlick A, Buszman P, Bochenek A, Schampaert E, Page P, Dressler O, Kosmidou I, Mehran R, Pocock SJ, Kappetein AP; EXCEL Trial Investigators. Everolimus-Eluting Stents or Bypass Surgery for Left Main Coronary Artery Disease. N Engl J Med. 2016 Dec 8;375(23):2223-2235. doi: 10.1056/NEJMoa1610227. Epub 2016 Oct 31. PMID 27797291
- [Derived] Farooq V, Serruys PW. Bypass Grafting Versus Percutaneous Intervention-Which Is Better in Multivessel Coronary Disease: Lessons From SYNTAX and Beyond. Prog Cardiovasc Dis. 2015 Nov-Dec;58(3):316-34. doi: 10.1016/j.pcad.2015.10.002. Epub 2015 Oct 31. PMID 26529569

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1905 subjects were randomized (Percutaneous Coronary Intervention (PCI): 948 & Coronary Artery Bypass Graft (CABG) 957) between September 29, 2010 and March 6, 2014. Five hundred and forty-nine (549) subjects were from 56 U.S. sites and 1356 subjects were from 70 international sites,for a total of 126 enrolling sites.
Pre-assignment Details: The original EXCEL study consisted of a randomized clinical trial (RCT) (n=2600) & a Universal Registry (n=1000). In February 2014,a decision was made to cap enrollment in the RCT at approximately 1900.The change in scope of the study design was not due to any device or subject safety issues.
Groups:
- Percutaneous Coronary Intervention (PCI): Those patients receiving the XIENCE PRIME™ EECSS or XIENCE V® EECSS or XIENCE Xpedition™ EECSS or XIENCE PRO EECSS
- Coronary Artery Bypass Graft (CABG): Those patients receiving Coronary Artery Bypass Graft (CABG)
Period: Overall Study
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Started | 948 | 957
Completed | 884 | 862
Not Completed | 64 | 95
Not completed — Lost to Follow-up | 53 | 61
Not completed — Withdrawal by Subject | 11 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG) | Total
Number analyzed (Participants) | 948 | 957 | 1905
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (9.6) | 65.9 (9.5) | 66.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 722 | 742 | 1464
  Male | 226 | 215 | 441
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 23 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 28 | 64
  White | 844 | 853 | 1697
  More than one race | 16 | 20 | 36
  Unknown or Not Reported | 31 | 33 | 64
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 534 | 541 | 1075
  United States | 278 | 271 | 549
  Canada | 103 | 100 | 203
  Southeast Asia | 7 | 8 | 15
  Australia | 6 | 9 | 15
  South America | 20 | 28 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: All deaths includes Cardiac death, Vascular death and Non-cardiovascular death.
  Myocardial Infarction (MI):
  * Q wave MI: Development of new, pathological Q wave on the ECG.
  * Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
  Stroke is defined as the rapid onset of a new persistent neurologic deficit attributed to an obstruction in cerebral blood flow and/or cerebral hemorrhage with no apparent non-vascular cause (e.g., trauma, tumor, or infection).
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 203 | 176

2. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 40 | 77

3. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 46 | 75
Statistical Analysis 1: Comparison: Percutaneous Coronary Intervention (PCI) vs Coronary Artery Bypass Graft (CABG); Test type: Non-Inferiority — p-value and 95% CI of the Difference derived from the Com-Nougue Approach of non-inferiority for two Kaplan-Meier Failure rates with a non-inferiority margin of 2% at the 0.05 level of significance; p < 0.0001, Com-Nougue — p-value and 95% CI of the Difference derived from the Com-Nougue Approach of non-inferiority for two Kaplan-Meier Failure rates with a non-inferiority margin of 2% at the 0.05 level of significance; Hazard Ratio (HR) = -3.1

4. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 66 | 97

5. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 80 | 106

6. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 115 | 122

7. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 137 | 135

8. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 173 | 154

9. Secondary Outcome: Number of Participants With All-cause Death, Protocol Defined MI or Protocol Defined Stroke
Description: as for outcome 1
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 203 | 176

10. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 1
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 40 | 82

11. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 1
Time Frame: 0 to 30 days
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 46 | 80

12. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 1
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 79 | 112

13. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 1
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 121 | 129

14. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 1
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 177 | 154

15. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: Death:
  * Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery).
  * Non-cardiac death is defined as a death not due to cardiac causes (as defined above).
  Myocardial Infarction (MI) -Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
  Unplanned revascularization for ischemia: Any repeat revascularization of either a target vessel or non-target vessel with any of the above criteria for ischemia met.
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 213 | 176
Statistical Analysis 1: Comparison: Percutaneous Coronary Intervention (PCI) vs Coronary Artery Bypass Graft (CABG); Test type: Non-Inferiority — p-value and 95% CI of the Difference derived from the Com-Nougue Approach of non-inferiority for two Kaplan-Meier Failure rates with a non-inferiority margin of 8.4% at the 0.05 level of significance; p = 0.011, Com-Nougue Approach — p-value and 95% CI of the Difference derived from the Com-Nougue Approach of non-inferiority for two Kaplan-Meier Failure rates with a non-inferiority margin of 8.4% at the 0.05 level of significance; Hazard Ratio (HR) = 4.0

16. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 15
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 260 | 203

17. Secondary Outcome: Number of Participants With Death, Protocol Defined MI, Protocol Defined Stroke or Unplanned Revascularization for Ischemia
Description: as for outcome 15
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 290 | 228

18. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  • Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  • Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  • Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 4 | 12

19. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 9 | 10

20. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 19 | 23

21. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 31 | 33

22. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 54 | 44

23. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 74 | 54

24. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 95 | 68

25. Secondary Outcome: Number of Participants With All-cause Mortality (Cardiac Death and Non-cardiac Death)
Description: as for outcome 18
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 119 | 89

26. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 34 | 58

27. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 37 | 59

28. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 46 | 68

29. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 53 | 68

30. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 64 | 73

31. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 74 | 78

32. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 86 | 81

33. Secondary Outcome: Number of Participants With Protocol Defined MI
Description: as for outcome 26
Time Frame: 0 to 5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 95 | 84

34. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: Stroke is defined as the rapid onset of a new persistent neurologic deficit attributed to an obstruction in cerebral blood flow and/or cerebral hemorrhage with no apparent non-vascular cause (e.g., trauma, tumor, or infection).
  Ischemic (Non-hemorrhagic): A stroke caused by an arterial obstruction due to either a thrombotic (e.g., large vessel disease/atherosclerotic or small vessel disease/lacunar) or embolic etiology.
  Hemorrhagic: A stroke due to a hemorrhage in the brain as documented by neuroimaging or autopsy. This category will include strokes due to primary intracerebral hemorrhage (intraparenchymal or intraventricular), ischemic strokes with hemorrhagic transformation (i.e., no evidence of hemorrhage on an initial imaging study but appearance on a subsequent scan), subdural hematoma,* and primary subarachnoid hemorrhage.
  * All subdural hematomas that develop during the clinical trial should be recorded and classified as either traumatic versus nontraumatic.
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 4 | 13

35. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 6 | 12

36. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 9 | 16

37. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 10 | 18

38. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 17 | 22

39. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 21 | 28

40. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 23 | 30

41. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke, and Hemorrhagic Stroke)
Description: as for outcome 34
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 26 | 33

42. Secondary Outcome: Number of Participants With Disability Following Stroke Event
Description: In case of an event of stroke disability at 90-days±2 weeks will be an overall measurement of severity of stroke as assessed by modified Rankin Scale (mRS) scale.
  Stroke disability will be classified using an adaptation of the modified Rankin Scale as follows, the assessment of which will be based on the Modified Rankin Disability Questionnaire.
  Scale 0; No stroke symptoms at all. (May have other complaints) Scale 1; No significant disability; symptoms present but no physical or other limitations.
  Scale 2; Slight disability; limitations in participation in usual social roles, but independent for activities of daily living (ADL) Scale 3; Some need for assistance but able to walk without assistance Scale 4; Moderately severe disability; need for assistance with some basic ADL, but not requiring constant care Scale 5; Severe disability; requiring constant nursing care and attention.
Time Frame: 90 days ± 2 weeks
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 17 | 29
Participants | 6 | 9

43. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations (TLR,TVR and Non-TVR)
Description: A target lesion (vessel) revascularization will be considered ischemia-driven if the target lesion diameter stenosis is ≥ 50% by QCA (analysis segment measurement, involving the lesion itself and 5 mm of proximal and/or distal margin) and any of the following criteria for ischemia are met:
  * A positive functional study corresponding to the area served by the target lesion; or
  * Ischemic ECG changes at rest in a distribution consistent with the target vessel; or
  * Typical ischemic symptoms referable to the target lesion; or
  * IVUS of the target lesion with a minimal lumen area (MLA) of ≤ 4 mm^2 for non left main lesions or ≤ 6 mm^2 for left main lesions. If the lesions are de novo (i.e. not restenotic), the
  * plaque burden must also be ≥ 60%; or
  * Fractional Flow Reserve (FFR) of the target lesion ≤ 0.80
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 3 | 12

44. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 6 | 13

45. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 28 | 29

46. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 62 | 40

47. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 95 | 56

48. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 114 | 67

49. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 4 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 143 | 81

50. Secondary Outcome: Number of Participants With Ischemia Driven Revascularizations
Description: as for outcome 43
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 150 | 88

51. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia-driven or Non Ischemia-driven)
Description: * A target lesion (vessel) revascularization will be considered ischemia-driven if the target lesion diameter stenosis is ≥ 50% by QCA (analysis segment measurement, involving the lesion itself and 5 mm of proximal and/or distal margin) and any of the following criteria for ischemia are met:
    * A positive functional study corresponding to the area served by the target lesion;
    * Ischemic ECG changes at rest in a distribution consistent with the target vessel;
    * Typical ischemic symptoms referable to the target lesion;
    * IVUS of the target lesion with a minimal lumen area (MLA) of ≤ 4 mm^2 for non left main lesions or ≤ 6 mm^2 for left main lesions. If the lesions are de novo (i.e. not restenotic), the
    * plaque burden must also be ≥ 60%;
    * FFR of the target lesion ≤ 0.80
  * A non target vessel revascularization will be considered ischemia-driven if any lesion the non target vessel has a diameter stenosis ≥ 50% by QCA with any of the above criteria for ischemia met.
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 3 | 12

52. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 7 | 13

53. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 29 | 30

54. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 63 | 42

55. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 97 | 57

56. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 116 | 68

57. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 146 | 83

58. Secondary Outcome: Number of Participants With All Revascularizations (Ischemia Driven and Not Ischemia Driven)
Description: as for outcome 51
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 153 | 92

59. Secondary Outcome: Percentage of Participants With Major Adverse Events (MAE)
Description: Composite of death, myocardial infarction, stroke, transfusion of ≥ 2 units of blood, major arrhythmia, unplanned coronary revascularization for ischemia, any unplanned surgery or radiologic procedure, renal failure, sternal wound dehiscence, infection requiring antibiotics for treatment, intubation for > 48 hours, or post-pericardiotomy syndrome.
Time Frame: In-hospital
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Percentage of participants
  Death | 0.4 | 1.3
  Myocardial infarction | 3.6 | 6.2
  Stroke | 0.4 | 1.4
  Transfusion of >= 2 units blood | 3.5 | 17.1
  TIMI major or minor bleeding | 3.0 | 9.3
  Major arrhythmia | 1.8 | 14.7
  Unplanned coronary revascularization for ischemia | 0.3 | 1.3
  Unplanned surgery/therapeutic radiologic procedure | 1.0 | 3.7
  Renal failure | 0.6 | 2.4
  Sternal wound dehiscence | 0.0 | 1.0
  Infection requiring antibiotics for treatment | 1.2 | 8.8
  Intubation for > 48 hours | 0.4 | 3.0
  Post-pericardiotomy syndrome | 0.0 | 0.2

60. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definition) Definite/Probable
Description: Definite stent thrombosis occurred by either angiographic/pathologic confirmation of stent thrombosis.
  Angiographic confirmation:The presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent&presence of at least 1 of the following criteria within a 48-hour time window:
  * Acute onset of ischemic symptoms at rest
  * New ischemic ECG changes
  * Typical rise&fall in cardiac biomarkers
  * Non-occlusive thrombus
  * Occlusive thrombus.
  Pathological confirmation: Evidence of recent thrombus within the stent determined at autopsy or via examination of tissue retrieved following thrombectomy.
  Probable stent thrombosis may occur after intracoronary stenting due to:
  * Unexplained death within first 30 days
  * Irrespective of the time after the index procedure,any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis&in the absence of any other obvious cause.
Time Frame: Early (0-30 days)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants
  Definite | 3 | 0
  Probable | 4 | 0

61. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definition) Definite/Probable
Description: as for outcome 60
Time Frame: Acute (<= 24 hours)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants
  Definite | 1 | 0
  Probable | 0 | 0

62. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definition) Definite/ Probable
Description: as for outcome 60
Time Frame: Subacute (1-30 days)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants
  Definite | 2 | 0
  Probable | 4 | 0

63. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definition) Definite/Probable
Description: as for outcome 60
Time Frame: Late (>30 days - 1 year)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants
  Definite | 0 | 0
  Probable | 1 | 0

64. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definition) Definite/ Probable
Description: as for outcome 60
Time Frame: Very late (>1 year)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants
  Definite | 3 | 0
  Probable | 1 | 0

65. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: Graft stenosis or occlusion is defined as Ischemic symptoms in the presence of ≥50% diameter stenosis in a coronary bypass graft.
Time Frame: In-hospital (≤ 7 days of index-procedure)
Population: ITT population. Subjects without the required follow-up are excluded from the time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 0 | 11

66. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 30 days
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 11

67. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 6 months
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 25

68. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 1 year
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 33

69. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 2 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 43

70. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 3 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 48

71. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 4 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 53

72. Secondary Outcome: Number of Participants With Graft Stenosis or Occlusion
Description: as for outcome 65
Time Frame: 0 to 5 years
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 0 | 58

73. Secondary Outcome: Number of Participants With Requirement for Blood Product Transfusion
Description: All TIMI definitions take into account blood transfusions, so that hemoglobin and hematocrit values are adjusted by 1 g/dl or 3%, respectively, for each unit of blood transfused. Therefore, the true change in hemoglobin or hematocrit if there has been an intervening transfusion between two blood measurements is calculated as follows:
  * Δ Hemoglobin = [baseline Hgb - post-transfusion Hgb] + [number of transfused units];
  * Δ Hematocrit = [baseline Hct - post-transfusion Hct] + [number of transfused units X 3].
Time Frame: 30 days
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 30 | 120

74. Secondary Outcome: Number of Participants With Requirement for Blood Product Transfusion
Description: as for outcome 73
Time Frame: 3 years
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 48 | 129

75. Secondary Outcome: Number of Participants With Requirement for Blood Product Transfusion
Description: as for outcome 73
Time Frame: 4 years
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 52 | 130

76. Secondary Outcome: Number of Participants With Requirement for Blood Product Transfusion
Description: as for outcome 73
Time Frame: 5 years
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 52 | 131

77. Secondary Outcome: Number of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding
Description: Bleeding will be classified by the TIMI hemorrhage classification
  Severity:
  Major:
  * Intracranial hemorrhage
  * A ≥5 g/dL decrease in the hemoglobin concentration
  * A ≥15% absolute decrease in the hematocrit
  Minor:
  * Observed blood loss:
    * A ≥ 3 g/dL decrease in the hemoglobin concentration
    * A ≥ 10% absolute decrease in the hematocrit
  * No observed blood loss:
    * A ≥ 4 g/dL decrease in the hemoglobin concentration
    * A ≥ 12% absolute decrease in the hematocrit
  Minimal:
  • Any clinically overt sign of hemorrhage (including imaging) that is associated with a < 3 g/dL decrease in hemoglobin concentration or < 9% decrease in the hematocrit.
Time Frame: 30 days
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 35 | 85

78. Secondary Outcome: Number of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding
Description: as for outcome 77
Time Frame: 3 years
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 114 | 132

79. Secondary Outcome: Number of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding
Description: as for outcome 77
Time Frame: 4 years
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 119 | 133

80. Secondary Outcome: Number of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major or Minor Bleeding
Description: as for outcome 77
Time Frame: 5 years
Population: ITT population. Analysis population includes subjects who had follow-up data at that time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 119 | 137

81. Secondary Outcome: Number of Participants With Bleeding Academic Research Consortium (BARC) Bleeding
Description: Type 0: No bleeding Type 1: Bleeding that is not actionable&does not cause the patient to seek unscheduled performance of studies,hospitalization,or treatment by a healthcare professional Type 2: Any overt, actionable sign of hemorrhage that does not fit the criteria for type 3,4,or 5 but does meet at least 1 of the following criteria:requiring nonsurgical, medical intervention by a healthcare professional; leading to hospitalization or increased level of care; prompting evaluation.
  Type 3 Type 3a
  * Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL
  * Any transfusion with overt bleeding Type 3b
  * Overt bleeding plus hemoglobin drop ≥5 g/dL*
  * Cardiac tamponade
  * Bleeding requiring surgical intervention for control
  * Bleeding requiring intravenous vasoactive agents Type 3c
  * Intracranial hemorrhage
  * Subcategories confirmed by autopsy or imaging or lumbar puncture
  * Intraocular bleed compromising vision Type 4: CABG-related bleeding Type 5: Fatal bleeding
Time Frame: 30 days
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 69 | 123

82. Secondary Outcome: Number of Participants With Bleeding Academic Research Consortium (BARC) Bleeding
Description: as for outcome 81
Time Frame: 3 years
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 109 | 145

83. Secondary Outcome: Number of Participants With Bleeding Academic Research Consortium (BARC) Bleeding
Description: as for outcome 81
Time Frame: 4 years
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 112 | 147

84. Secondary Outcome: Number of Participants With Bleeding Academic Research Consortium (BARC) Bleeding
Description: as for outcome 81
Time Frame: 5 years
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 113 | 153

85. Secondary Outcome: Number of Participants With Major Adverse Events (MAE)
Description: * death
  * myocardial infarction
  * stroke
  * Transfusion of ≥2 units of blood
  * TIMI major or minor bleeding
  * major arrhythmia
  * unplanned coronary revascularization for ischemia
  * any unplanned surgery or therapeutic radiologic procedure
  * renal failure
  * sternal wound dehiscence
  * infection requiring antibiotics for treatment
  * intubation for > 48 hours
  * post-pericardiotomy syndrome
Time Frame: 30 days
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants
  Death | 9 | 10
  Myocardial infarction | 37 | 59
  Stroke | 6 | 12
  Transfusion of >= 2 units blood | 38 | 163
  TIMI major or minor bleeding | 35 | 85
  Major arrhythmia | 20 | 154
  Unplanned coronary revascularization for ischemia | 6 | 13
  Unplanned surgery/therapeutic radiologic procedure | 12 | 39
  Renal failure | 6 | 24
  Sternal wound dehiscence | 0 | 19
  Infection requiring antibiotics for treatment | 24 | 133
  Intubation for > 48 hours | 4 | 28
  Post-pericardiotomy syndrome | 0 | 4

86. Secondary Outcome: Number of Participants With Complete Revascularization (Residual = 0)
Description: 1. Complete anatomic revascularization requires revascularization of all vessels ≥2.0 mm reference vessel diameter with a DS ≥60% (both as measured by core angiographic laboratory analysis).
     -While this will be the pre-specified criteria for anatomically significant lesions, sensitivity analysis will be performed using different criteria (e.g. ≥2.5 mm vessels, DS ≥70%, etc.)
  2. From the baseline angiogram, the angiographic core lab will identify and designate those lesions and vessels requiring revascularization in all subjects according to this definition, prior to knowledge of the extent of actual revascularization.
  3. Following PCI, the angiographic core lab will determine the extent of revascularization (vessels with TIMI 2or3 flow post procedure with a core laboratory DS <50% considered successfully revascularized).
  4. Following CABG, the angiographic core lab will determine the extent of revascularization or if there is a repeat angiogram during the index hospitalization.
Time Frame: At Baseline
Population: Not all PCI patients have Baseline and Post-PCI Syntax score assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 917 | 21
Participants | 259 | 10

87. Secondary Outcome: Number of Participants With Definite Stent Thrombosis (ST) or Symptomatic Graft Occlusion
Description: - Definite ST occurred by either angiographic/pathologic confirmation of ST.
  Angiographic confirmation:The presence of a thrombus that originates in the stent/in the segment 5mm proximal/distal to the stent&presence of at least 1 of the following criteria within 48-hours:
  * Acute onset of ischemic symptoms at rest
  * New ischemic ECG changes
  * Typical rise&fall in cardiac biomarkers
  * Non-occlusive &occlusive thrombus
  Pathological confirmation:Evidence of recent thrombus within the stent determined at autopsy/via examination of tissue retrieved following thrombectomy.
  -Symptomatic graft occlusion: Ischemic symptoms in the presence of ≥50% diameter stenosis in a coronary bypass graft.
Time Frame: In-hospital (≤ 7 days of post index procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 942 | 940
Participants | 1 | 11

88. Secondary Outcome: Number of Participants With Definite Stent Thrombosis or Symptomatic Graft Occlusion
Description: as for outcome 87
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 3 | 33

89. Secondary Outcome: Number of Participants With Definite Stent Thrombosis or Symptomatic Graft Occlusion
Description: as for outcome 87
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 5 | 43

90. Secondary Outcome: Number of Participants With Definite Stent Thrombosis or Symptomatic Graft Occlusion
Description: as for outcome 87
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 7 | 48

91. Secondary Outcome: Number of Participants With Definite Stent Thrombosis or Symptomatic Graft Occlusion
Description: as for outcome 87
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 10 | 53

92. Secondary Outcome: Number of Participants With Definite Stent Thrombosis or Symptomatic Graft Occlusion
Description: as for outcome 87
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
Number analyzed (Participants) | 948 | 957
Participants | 10 | 58

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Percutaneous Coronary Intervention (PCI) | Coronary Artery Bypass Graft (CABG)
All-Cause Mortality (participants affected / at risk) | 119/948 | 89/957
Serious Adverse Events (participants affected / at risk) | 535/948 | 550/957
Other Adverse Events (participants affected / at risk) | 791/948 | 831/957
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Percutaneous Coronary Intervention (PCI) (N=948) | Coronary Artery Bypass Graft (CABG) (N=957)
Anemia (Blood and lymphatic system disorders) | 18 | 9
Bleeding (Blood and lymphatic system disorders) | 31 | 40
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Epistaxis (Blood and lymphatic system disorders) | 2 | 1
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 24 | 10
Other (Blood and lymphatic system disorders) | 12 | 12
Respiratory tract bleeding (Blood and lymphatic system disorders) | 1 | 1
Retroperitoneal bleeding (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Abrupt closure (Cardiac disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 21 | 13
Angina pectoris (includes atypical angina and cardiac chest pain) (Cardiac disorders) | 100 | 54
Angina unstable (Cardiac disorders) | 31 | 17
Asystole (Cardiac disorders) | 2 | 6
Atrial fibrillation (Cardiac disorders) | 26 | 36
Atrial flutter (Cardiac disorders) | 4 | 8
Bradycardia (Cardiac disorders) | 6 | 8
Cardiac : Other (Cardiac disorders) | 53 | 36
Cardiac arrest (Cardiac disorders) | 10 | 6
Cardiac enzymes increased (Cardiac disorders) | 5 | 4
Cardiac functional test abnormal (Cardiac disorders) | 6 | 2
Cardiac tamponade (Cardiac disorders) | 5 | 4
Cardiac valve disorder/disease (Cardiac disorders) | 4 | 4
Cardio-respiratory arrest (Cardiac disorders) | 4 | 3
Cardiogenic shock (Cardiac disorders) | 5 | 9
Cardiomyopathy (Cardiac disorders) | 2 | 2
Conduction disorder (including AV block, BBB) (Cardiac disorders) | 3 | 9
Congestive heart failure (Cardiac disorders) | 31 | 37
Coronary arteriospasm (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 8 | 0
Coronary artery graft occlusion (Cardiac disorders) | 1 | 30
Coronary artery in-stent restenosis (Cardiac disorders) | 26 | 2
Coronary artery occlusion (Cardiac disorders) | 3 | 6
Coronary artery perforation (Cardiac disorders) | 1 | 0
Coronary artery reocclusion (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 19 | 7
Coronary stent thrombosis (Cardiac disorders) | 7 | 1
Hypertension (Cardiac disorders) | 3 | 2
Hypertensive crisis (Cardiac disorders) | 3 | 2
Hypotension (Cardiac disorders) | 9 | 3
Myocardial infarction (Cardiac disorders) | 73 | 47
No-reflow phenomenon/slow flow (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 5
Pericardial effusion (Cardiac disorders) | 2 | 4
Plaque shift (tissue breakdown associated with device) (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 0
Ventricular fibrillation (Cardiac disorders) | 7 | 4
Ventricular tachycardia (sustained) (Cardiac disorders) | 1 | 7
electrocardiogram (ECG) abnormal (Cardiac disorders) | 3 | 1
Diabetes mellitus (Endocrine disorders) | 5 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Other : Endocrine disorder (Endocrine disorders) | 4 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Colonic/intestinal polyp (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Dysphagia (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastroenteritis (Gastrointestinal disorders) | 3 | 1
Gastroesophageal reflux diseases (Gastrointestinal disorders) | 1 | 2
Gastrointestinal ulcer/peptic ulcer (Gastrointestinal disorders) | 6 | 3
Hepatobiliary disease (Gastrointestinal disorders) | 8 | 8
Intestinal obstruction (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 0 | 2
Other : Gastrointestinal disorder (Gastrointestinal disorders) | 27 | 29
Pancreatic disorder (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 5
Accidents (General disorders) | 0 | 1
Cataract (General disorders) | 1 | 1
Chest pain (non-cardiac or non-specific) (General disorders) | 10 | 4
Dehydration (General disorders) | 3 | 2
Edema peripheral (General disorders) | 1 | 1
Eye disorders (General disorders) | 1 | 1
Fall (General disorders) | 4 | 0
Fatigue/Weakness (General disorders) | 2 | 3
Fever/Pyrexia (General disorders) | 1 | 2
Headache (General disorders) | 0 | 1
Injury (General disorders) | 1 | 1
Other (General disorders) | 11 | 15
Other shock (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Allergic conditions : Other (Immune system disorders) | 0 | 1
Contrast media allergy/reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity/drug allergy (Immune system disorders) | 0 | 1
Hypersensitivity/allergic reaction (Immune system disorders) | 1 | 3
Bone and joint infections (Infections and infestations) | 5 | 6
Cellulitis (Infections and infestations) | 6 | 5
Deep sternal wound infection (Infections and infestations) | 1 | 14
Flu/influenza (Infections and infestations) | 3 | 0
Gastrointestinal infection (Infections and infestations) | 4 | 4
Genitourinary infection (Infections and infestations) | 8 | 11
Lower respiratory tract infection (Infections and infestations) | 7 | 16
Other : Infection (Infections and infestations) | 25 | 26
Skin and subcutaneous infection (Infections and infestations) | 6 | 11
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Vein harvest site infection (Infections and infestations) | 1 | 6
Catheter site hematoma (Injury, poisoning and procedural complications) | 2 | 0 — Percutaneous coronary intervention (PCI) complications: access site complications
Other : Percutaneous coronary intervention (PCI) complications (Injury, poisoning and procedural complications) | 4 | 2 — Percutaneous coronary intervention (PCI) complications: access site complications
Blood creatinine increased (Investigations) | 3 | 3
Elevated cardiac enzymes (Investigations) | 8 | 3
Hemoglobin decreased (Investigations) | 7 | 2
Hyperglycaemia (Investigations) | 3 | 2
Hyperkalemia (Investigations) | 4 | 2
Hypoglycemia (Investigations) | 1 | 0
Hypokalemia (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 0 | 1
Other (Investigations) | 2 | 5
Other abnormal blood test (Investigations) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Backpain (Musculoskeletal and connective tissue disorders) | 3 | 2
Fracture (Musculoskeletal and connective tissue disorders) | 10 | 21
Joint or tendon disease/disorder (Musculoskeletal and connective tissue disorders) | 6 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Other : Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 10 | 12
Spinal disorder (Musculoskeletal and connective tissue disorders) | 5 | 2
Neoplasm/cancer : Blood or lymphatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Neoplasm/cancer : Gastrointestinal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 4
Neoplasm/cancer : Musculoskeletal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neoplasm/cancer : Nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm/cancer : Reproductive system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neoplasm/cancer : Respiratory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 6
Neoplasm/cancer : Skin or subcutaneous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Neoplasm/cancer : Urinary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Other :Neoplasm/cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 14
Cerebrovascular accident (CVA) (Nervous system disorders) | 27 | 36
Dizziness (Nervous system disorders) | 4 | 2
Encephalopathy (Nervous system disorders) | 1 | 1
Other : Neurological/psychiatric disorders (Nervous system disorders) | 9 | 13
Seizure/convulsion (Nervous system disorders) | 3 | 3
Syncope/fainting/loss of consciousness (Nervous system disorders) | 2 | 2
Transient ischemic attack (TIA) (Nervous system disorders) | 6 | 11
Vertigo (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Mental status change (Psychiatric disorders) | 1 | 0
Psychiatric disorder (Psychiatric disorders) | 2 | 1
Benign prostatic hyperplasia (Renal and urinary disorders) | 4 | 3
Incontinence (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 3
Other : Renal and urinary disorder (Renal and urinary disorders) | 14 | 10
Renal artery stenosis (Renal and urinary disorders) | 0 | 3
Renal failure (Renal and urinary disorders) | 17 | 14
Renal insufficiency/impairment (Renal and urinary disorders) | 7 | 17
Urinary retention (Renal and urinary disorders) | 1 | 3
Urinary stone/calculus (Renal and urinary disorders) | 2 | 4
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
COPD (chronic obstructive pulmonary disease) (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 13 | 14
Other : Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 19 | 30
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 27
Aneurysm (Vascular disorders) | 2 | 2
Claudication (Vascular disorders) | 8 | 6
Deep vein thrombosis (Vascular disorders) | 3 | 4
Dissection (Vascular disorders) | 3 | 4
Embolism (Vascular disorders) | 0 | 1
Other : Peripheral vascular disorder (Vascular disorders) | 4 | 5
Peripheral artery disease/peripheral venous disease (Vascular disorders) | 13 | 19
Peripheral nerve lesion/injury (including peripheral neuropathy) (Vascular disorders) | 0 | 1
Pseudoaneurysm (Vascular disorders) | 2 | 3
Stenosis (Vascular disorders) | 6 | 10
Thrombosis (non stent/non-coronary) (Vascular disorders) | 2 | 3
Vascular occlusion (Vascular disorders) | 4 | 6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Percutaneous Coronary Intervention (PCI) (N=948) | Coronary Artery Bypass Graft (CABG) (N=957)
Anemia (Blood and lymphatic system disorders) | 42 | 83
Bleeding (Blood and lymphatic system disorders) | 75 | 121
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Epistaxis (Blood and lymphatic system disorders) | 10 | 7
Gastrointestinal bleeding (Blood and lymphatic system disorders) | 36 | 15
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Other (Blood and lymphatic system disorders) | 47 | 33
Respiratory tract bleeding (Blood and lymphatic system disorders) | 2 | 1
Retroperitoneal bleeding (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 16
Abrupt closure (Cardiac disorders) | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 21 | 14
Angina pectoris (includes atypical angina and cardiac chest pain) (Cardiac disorders) | 205 | 124
Angina unstable (Cardiac disorders) | 42 | 22
Asystole (Cardiac disorders) | 2 | 7
Atrial fibrillation (Cardiac disorders) | 54 | 201
Atrial flutter (Cardiac disorders) | 7 | 17
Bradycardia (Cardiac disorders) | 24 | 25
Cardiac arrest (Cardiac disorders) | 10 | 7
Cardiac enzymes increased (Cardiac disorders) | 16 | 18
Cardiac functional test abnormal (Cardiac disorders) | 6 | 2
Cardiac tamponade (Cardiac disorders) | 5 | 4
Cardiac valve disorder/disease (Cardiac disorders) | 4 | 6
Cardio-respiratory arrest (Cardiac disorders) | 4 | 3
Cardiogenic shock (Cardiac disorders) | 5 | 10
Cardiomyopathy (Cardiac disorders) | 4 | 6
Conduction disorder (including atrioventricular block (AV block, bundle branch block(BBB)) (Cardiac disorders) | 6 | 16
Congestive heart failure (Cardiac disorders) | 39 | 50
Coronary arteriospasm (Cardiac disorders) | 0 | 2
Coronary artery dissection (Cardiac disorders) | 23 | 1
Coronary artery embolism (Cardiac disorders) | 0 | 0
Coronary artery graft occlusion (Cardiac disorders) | 1 | 34
Coronary artery in-stent restenosis (Cardiac disorders) | 27 | 3
Coronary artery occlusion (Cardiac disorders) | 7 | 6
Coronary artery perforation (Cardiac disorders) | 3 | 1
Coronary artery reocclusion (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 20 | 8
Coronary stent thrombosis (Cardiac disorders) | 7 | 2
Electrocardiogram (ECG) abnormal (Cardiac disorders) | 10 | 14
Hypertension (Cardiac disorders) | 31 | 42
Hypertensive crisis (Cardiac disorders) | 4 | 4
Hypotension (Cardiac disorders) | 32 | 23
Myocardial infarction (Cardiac disorders) | 78 | 58
No-reflow phenomenon/slow flow (Cardiac disorders) | 9 | 0
Other (Cardiac disorders) | 103 | 85
Palpitations (Cardiac disorders) | 12 | 16
Pericardial effusion (Cardiac disorders) | 4 | 11
Plaque shift (tissue breakdown associated with device) (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 12 | 18
Ventricular fibrillation (Cardiac disorders) | 7 | 5
Ventricular tachycardia (sustained) (Cardiac disorders) | 4 | 8
Diabetes mellitus (Endocrine disorders) | 21 | 19
Hyperthyroidism (Endocrine disorders) | 0 | 3
Hypothyroidism (Endocrine disorders) | 6 | 5
Other (Endocrine disorders) | 9 | 18
Abdominal discomfort (Gastrointestinal disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 16 | 14
Colonic/intestinal polyp (Gastrointestinal disorders) | 12 | 5
Constipation (Gastrointestinal disorders) | 9 | 13
Diarrhoea (Gastrointestinal disorders) | 18 | 19
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 2
Gastritis (Gastrointestinal disorders) | 4 | 11
Gastroenteritis (Gastrointestinal disorders) | 5 | 5
Gastrointestinal ulcer/peptic ulcer (Gastrointestinal disorders) | 8 | 3
Gastrooesophageal reflux diseases (Gastrointestinal disorders) | 12 | 12
Hepatobiliary disease (Gastrointestinal disorders) | 11 | 13
Intestinal obstruction (Gastrointestinal disorders) | 4 | 5
Nausea (Gastrointestinal disorders) | 7 | 20
Other (Gastrointestinal disorders) | 69 | 61
Pancreatic disorder (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 12 | 17
Accidents (General disorders) | 0 | 2
Cataract (General disorders) | 4 | 8
Chest pain (non-cardiac or non-specific) (General disorders) | 30 | 26
Dehydration (General disorders) | 3 | 4
Ear disorders (General disorders) | 3 | 2
Ecchymosis (General disorders) | 4 | 1
Edema peripheral (General disorders) | 15 | 17
Eye disorders (General disorders) | 3 | 9
Fall (General disorders) | 10 | 2
Fatigue/Weakness (General disorders) | 20 | 25
Fever/Pyrexia (General disorders) | 4 | 6
Headache (General disorders) | 6 | 3
Injury (General disorders) | 4 | 4
Other (General disorders) | 53 | 56
Other shock (General disorders) | 0 | 1
Pain (General disorders) | 6 | 8
Pruritis (General disorders) | 0 | 1
Rash (General disorders) | 5 | 6
Allergy to metal (Immune system disorders) | 0 | 1
Contrast media allergy/reaction (Immune system disorders) | 4 | 0
Drug hypersensitivity/drug allergy (Immune system disorders) | 19 | 11
Hypersensitivity/allergic reaction (Immune system disorders) | 11 | 5
Other (Immune system disorders) | 8 | 7
Bone and joint infections (Infections and infestations) | 7 | 6
Cellulitis (Infections and infestations) | 12 | 11
Deep sternal wound infection (Infections and infestations) | 1 | 18
Flu/influenza (Infections and infestations) | 5 | 2
Gastrointestinal infection (Infections and infestations) | 6 | 9
Genitourinary infection (Infections and infestations) | 25 | 43
Joint infection (Infections and infestations) | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 28 | 57
Other (Infections and infestations) | 43 | 61
Skin and subcutaneous infection (Infections and infestations) | 14 | 34
Upper respiratory tract infection (Infections and infestations) | 26 | 25
Vein harvest site infection (Infections and infestations) | 1 | 19
Catheter site hematoma (Injury, poisoning and procedural complications) | 24 | 1 — Percutaneous coronary intervention (PCI) complications: access site complications
Catheter site pain (Injury, poisoning and procedural complications) | 3 | 0 — Percutaneous coronary intervention (PCI) complications: access site complications
Catheter site swelling (Injury, poisoning and procedural complications) | 1 | 0 — Percutaneous coronary intervention (PCI) complications: access site complications
Cathether site bleeding (Injury, poisoning and procedural complications) | 4 | 0 — Percutaneous coronary intervention (PCI) complications: access site complications
Other (Injury, poisoning and procedural complications) | 12 | 2 — Percutaneous coronary intervention (PCI) complications: access site complications
Blood creatinine increased (Investigations) | 12 | 11
Blood creatinine phosphokinase increased (Investigations) | 0 | 1
Elevated cardiac enzymes (Investigations) | 44 | 88
Hematocrit decreased (Investigations) | 1 | 5
Hemoglobin decreased (Investigations) | 17 | 35
Hyperglycaemia (Investigations) | 3 | 16
Hyperkalaemia (Investigations) | 7 | 9
Hyperlipidaemia/hypercholesterolemia (Investigations) | 5 | 4
Hypoglycemia (Investigations) | 1 | 2
Hypokalaemia (Investigations) | 9 | 11
Liver function test abnormal (Investigations) | 8 | 14
Other (Investigations) | 14 | 37
Other abnormal blood test (Investigations) | 4 | 16
Arthritis (Musculoskeletal and connective tissue disorders) | 20 | 16
Backpain (Musculoskeletal and connective tissue disorders) | 24 | 23
Fracture (Musculoskeletal and connective tissue disorders) | 22 | 30
Joint or tendon disease/disorder (Musculoskeletal and connective tissue disorders) | 21 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 49 | 60
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 6
Other (Musculoskeletal and connective tissue disorders) | 69 | 69
Spinal disorder (Musculoskeletal and connective tissue disorders) | 9 | 8
Neoplasm/cancer : Blood or lymphatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Neoplasm/cancer : Gastrointestinal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 5
Neoplasm/cancer : Musculoskeletal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neoplasm/cancer : Nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm/cancer : Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 16
Neoplasm/cancer : Reproductive system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Neoplasm/cancer : Respiratory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 6
Neoplasm/cancer : Skin or subcutaneous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 11
Neoplasm/cancer : Urinary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10
Cerebrovascular accident (CVA) (Nervous system disorders) | 29 | 36
Dizziness (Nervous system disorders) | 11 | 9
Encephalopathy (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 1 | 3
Other : Neurological/psychiatric disorders (Nervous system disorders) | 28 | 51
Seizure/convulsion (Nervous system disorders) | 3 | 6
Sleep disorder (Nervous system disorders) | 0 | 3
Syncope/fainting/loss of consciousness (Nervous system disorders) | 9 | 6
Transient ischemic attack (TIA) (Nervous system disorders) | 10 | 18
Vertigo (Nervous system disorders) | 3 | 4
Agitation (Psychiatric disorders) | 1 | 6
Anxiety (Psychiatric disorders) | 5 | 8
Confusion (Psychiatric disorders) | 4 | 7
Dementia (Psychiatric disorders) | 1 | 3
Depression (Psychiatric disorders) | 9 | 9
Mental status change (including coma) (Psychiatric disorders) | 3 | 1
Psychiatric disorder (Psychiatric disorders) | 2 | 2
Benign prostatic hyperplasia (Renal and urinary disorders) | 10 | 7
Incontinence (Renal and urinary disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 3 | 3
Other (Renal and urinary disorders) | 32 | 40
Renal artery stenosis (Renal and urinary disorders) | 1 | 3
Renal failure (Renal and urinary disorders) | 21 | 24
Renal insufficiency/impairment (Renal and urinary disorders) | 20 | 28
Urinary retention (Renal and urinary disorders) | 8 | 6
Urinary stone/calculus (Renal and urinary disorders) | 6 | 9
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 4
COPD (chronic obstructive pulmonary disease) (Respiratory, thoracic and mediastinal disorders) | 23 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Dyspnea/shortness of breath (Respiratory, thoracic and mediastinal disorders) | 58 | 57
Other (Respiratory, thoracic and mediastinal disorders) | 51 | 101
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 63
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 18 | 14
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 38
Aneurysm (Vascular disorders) | 4 | 6
Arteriovenous fistula (Vascular disorders) | 0 | 1
Claudication (Vascular disorders) | 12 | 16
Deep vein thrombosis (Vascular disorders) | 5 | 7
Embolism (Vascular disorders) | 0 | 1
Other (Vascular disorders) | 14 | 19
Peripheral artery disease/peripheral venous disease (Vascular disorders) | 26 | 27
Peripheral nerve lesion/injury (Vascular disorders) | 2 | 2
Pseudoaneurysm (Vascular disorders) | 2 | 4
Stenosis (Vascular disorders) | 17 | 11
Thrombophlebitis (Vascular disorders) | 3 | 4
Thrombosis (non stent/non-coronary) (Vascular disorders) | 2 | 4
Vascular occlusion (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT01205776/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT01205776/SAP_001.pdf